CLINICAL TRIAL: NCT01947894
Title: SWEGHO - A PROSPECTIVE NON INTERVENTIONAL STUDY PROTOCOL WITH PRIMARY DATA COLLECTION - ASSESSMENT OF THE LONG TERM TREATMENT OUTCOMES OF GENOTROPIN TREATMENT IN GHD PATIENTS IN SWEDEN
Brief Title: A Prospective Non-Interventional Study Protocol With Primary Data Collection - Assessment Of The Long Term Treatment Outcomes Of Genotropin Treatment In Growth Hormone Deficiency (GHD) Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6281313; SWEGHO (Other: Alias Study Number)
Record Dates: First submitted 2013-06-18; First posted 2013-09-23 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Growth Hormone deficient Patients: Patients with GHD on Genotropin® replacement therapy.
  Interventions: Other: Non Interventional Study

INTERVENTIONS:
Other: Non Interventional Study — Non Interventional Study

SUMMARY:
The purpose of this study is to assess the long term treatment outcomes of Growth Hormone treatment in patients who are prescribed and treated with Genotropin. Also, plan to determine the relationships between clinical status, dosage schedule and response to Genotropin treatment.

This study will also contribute to our knowledge of adult Growth Hormone Deficiency, including transition period in Childhood Onset Growth Hormone Deficiency and its treatment.

DETAILED DESCRIPTION:
Patients within inclusion criteria are asked to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of 18 years of age and above and fulfilling one of the three alternatives a-c below;

  1. Newly diagnosed with GHD according to the current medical standard.
  2. Diagnosed with GHD before 2013 and previously treated with Genotropin and followed in KIMS®.
  3. Transition patients diagnosed with CO-GHD before 2013.
* Prescribed Genotropin at the time of inclusion.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients who participate in any concurrent clinical interventional trial where a non-authorized or authorized study medication is used, during their participation in Swedish KIMS® Xtended. Concurrent studies which do not include any study interventional items (whether medications or devices) are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients wiht Growth Hormone Deficiency
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2013-11-20 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Sweden (12):
  - Vastra Gotalands Regionen, Skövde, Skaraborg
  - Landstinget Dalarna, Falun
  - Sahlgrenska University hospital, Gothenburg
  - Central Hospital/ Department of Medicine, Kristianstad
  - Universitetssjukhuset, EM-kliniken, Linköping
  - Ljungby Lasarettet, Ljungby
  - University Hospital SUS, Malmo
  - Landstinget i Stockholms Lan, Stockholm
  - Karolinska Universitetssjukhuset, Kliniken for Endokrinologi, Stockholm
  - Akademiska sjukhuset / Medicincentrum, Diabetes- och Endokrinsektionen, Uppsala
  - Medicinkliniken, Centrallasarettet Vaxjo, Vaxjo
  - Landstinget i Jonkopings Lan, Värnamo

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281313&StudyName=A%20Prospective%20Non-Interventional%20Study%20Protocol%20With%20Primary%20Data%20Collection%20-%20%20Assessment%20Of%20The%20Long%20Term%20Treatment%20Outcomes%20Of%20Genotr

RESULTS

PARTICIPANT FLOW:
Groups:
- KIMS Adult Onset Growth Hormone Deficiency (GHD): Participants were diagnosed with GHD before 2013, were previously treated with Genotropin and were followed in KIMS®. Participants continued to be diagnosed with GHD as per current medical standards, who aged greater than or equal to (>=) 18 years, received Genotropin treatment in a real world clinic setting as prescribed in clinical practice and were followed up/observed for long-term Genotropin therapy treatment outcomes in this study. KIMS® (Pfizer international metabolic database), have data for long-term safety and treatment outcomes of adult participants treated with Genotropin in a real-world clinical setting between 1994 and 2012.
- Naive Adult Onset GHD: Participants who were newly diagnosed with GHD as per current medical standards, aged >=18 years, received Genotropin treatment in a real world clinic setting as prescribed in clinical practice and were followed up/observed for long-term Genotropin therapy treatment outcomes in this study.
- Childhood Onset Growth Hormone Deficiency (CO-GHD): Participants were diagnosed with CO-GHD before 2013. Participants aged >=18 years and continued to be diagnosed with GHD as per current medical standards, received Genotropin treatment in a real world clinic setting as prescribed in clinical practice and were followed up/observed for long-term Genotropin therapy treatment outcomes in this study.
Period: Overall Study
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Started | 247 | 42 | 88
Treated | 246 | 41 | 87
Completed | 160 | 24 | 61
Not Completed | 87 | 18 | 27
Not completed — Other | 3 | 4 | 3
Not completed — Withdrawal by Subject | 12 | 4 | 1
Not completed — Death | 12 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Adverse Event | 5 | 1 | 0
Not completed — Switched to other growth hormone brand | 53 | 8 | 23

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD) | Total
Number analyzed (Participants) | 247 | 42 | 88 | 377
Age, Customized [Count of Participants; unit: Participants]
  0 to less than or equal to (<=) 18 Years | 0 | 0 | 0 | 0
  Greater than (>) 18 to less than (<) 65 Years | 138 | 38 | 83 | 259
  >=65 Years | 100 | 4 | 2 | 106
  Unknown | 9 | 0 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 22 | 42 | 184
  Male | 127 | 20 | 46 | 193
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified According to Insulin-like Growth Factor (IGF-I) Assessments
Description: IGF-I along with growth hormone helps promote normal bone and tissue growth and development. Categories for assessment for participant's post-baseline IGF-I values: (1) IGF-I LLN = if any of assessments of IGF-I post-baseline visit was lower than lower limit of normal (LLN); (2) IGF-I ULN = If any of assessments of IGF-I post-baseline visit was greater than upper level of normal (ULN); (3) IGF-I unknown = no IGF-I reported; (4) Within reference range = IGF-I levels within normal range. Following is normal reference range of IGF-I in nanogram per milliliter. 18 Years of age (Y): Male =162-541, Female =170-640; 19 Y: Male =138-442, Female =147-527; 20 Y: Male =122-384,Female =132-457; 21-25 Y=116-341; 26-30 Y=117-321; 31-35 Y=113-297; 36-40 Y=106-277; 41-45 Y =98-261; 46-50 Y=91-246; 51-55 Y=84-233; 56-60 Y=78-220; 61-65 Y=72-207; 66-70 Y=67-195; 71-75 Y=62-184; 76-80 Y=57-172; >80 Y=53-162. There was no differentiation for male and female in normal range of IGF-I after 20 years of age.
Time Frame: Up to 5 years (after baseline visit)
Population: Full analysis set (FAS) included all correctly enrolled participants who received at least 1 dose of Genotropin. Erroneously enrolled participants were excluded from FAS, as they did not meet the inclusion criteria or met an exclusion criterion, which was discovered after enrolment to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
Participants
  IGF-I LLN | 11 | 2 | 4
  IGF-I ULN | 63 | 8 | 30
  IGF-I ULN within reference range | 159 | 22 | 47
  IGF-I Unknown | 13 | 6 | 6

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received Genotropin without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 5 years
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Genotropin.
Measure: Count of Participants; unit: Participants
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 41 | 87
Participants
  AEs | 103 | 17 | 22
  SAEs | 57 | 5 | 10

3. Secondary Outcome: Number of Treatment Related Adverse Events
Description: Treatment-related AEs refer to AEs that have a causal relationship with the treatment or usage. If there was any relationship between AE and Genotropin treatment,that was judged by investigator.
Time Frame: Baseline up to 5 years
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Genotropin. "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure.
Measure: Number; unit: adverse events
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 103 | 17 | 22
adverse events | 8 | 2 | 0

4. Secondary Outcome: Number of Adverse Events Leading to Withdrawal of Genotropin Treatment
Description: An AE is any untoward medical occurrence in a participant administered a medicinal product that need not necessarily have a causal relationship with the product treatment or usage. An SAE is any untoward medical occurrence in a participant administered a medicinal or nutritional product at any dose that resulted to death, life-threatening, hospitalization or prolongation of hospitalization, persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); and congenital anomaly/birth defect.
Time Frame: Baseline up to 5 years
Population: as for outcome 3
Measure: Number; unit: adverse events
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 103 | 117 | 22
adverse events | 14 | 2 | 1

5. Secondary Outcome: Number of Participants Who Discontinued Study Due to Adverse Events
Description: An AE is any untoward medical occurrence in a participant administered a medicinal product that need not necessarily have a causal relationship with the product treatment or usage. An SAE is any untoward medical occurrence in a participant administered a medicinal or nutritional product at any dose that resulted to death, life-threatening, hospitalization or prolongation of hospitalization, persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); and congenital anomaly/birth defect. Participants who discontinued study due to AEs were reported.
Time Frame: Baseline up to 5 years
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Genotropin.
Measure: Count of Participants; unit: Participants
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 41 | 87
Participants | 5 | 1 | 0

6. Secondary Outcome: Weight of Participants at Baseline, Years 1, 2, 3, 4 and 5
Description: Weight of participants was measured in kilograms (kg).
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: FAS was analyzed. Here, "Number analyzed" = participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
kg
  Baseline: number analyzed (Participants) | 232 | 33 | 81
  Baseline | 83.8 (16.76) | 82.4 (19.68) | 86.9 (26.11)
  Year 1: number analyzed (Participants) | 168 | 20 | 51
  Year 1 | 83.9 (18.09) | 86.4 (15.54) | 84.3 (25.11)
  Year 2: number analyzed (Participants) | 156 | 21 | 45
  Year 2 | 82.8 (15.66) | 86.8 (15.54) | 87.7 (20.73)
  Year 3: number analyzed (Participants) | 103 | 14 | 45
  Year 3 | 85.4 (18.91) | 84.3 (17.67) | 89.4 (24.08)
  Year 4: number analyzed (Participants) | 70 | 5 | 27
  Year 4 | 82.4 (17.83) | 97.2 (9.20) | 82.5 (20.66)
  Year 5: number analyzed (Participants) | 11 | 0 | 2
  Year 5 | 79.5 (16.00) |  | 104.4 (0.85)

7. Secondary Outcome: Change From Baseline in Weight of Participants at Years 1, 2, 3, 4 and 5
Description: Weight of participants was measured in kg.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
kg
  Change at Year 1: number analyzed (Participants) | 162 | 18 | 49
  Change at Year 1 | 0 (6.55) | -2.0 (15.37) | -2.3 (21.49)
  Change at Year 2: number analyzed (Participants) | 150 | 18 | 45
  Change at Year 2 | -0.7 (6.82) | -1.6 (12.85) | 1.0 (5.65)
  Change at Year 3: number analyzed (Participants) | 98 | 14 | 40
  Change at Year 3 | 2.2 (11.41) | -0.3 (13.41) | -2.8 (18.16)
  Change at Year 4: number analyzed (Participants) | 67 | 5 | 26
  Change at Year 4 | -1.6 (8.44) | 6.6 (7.24) | -0.3 (7.52)
  Change at Year 5: number analyzed (Participants) | 11 | 0 | 2
  Change at Year 5 | -2.2 (8.02) |  | -12.9 (20.22)

8. Secondary Outcome: Height of Participants at Baseline, Years 1, 2, 3, 4 and 5
Description: Height of participants was measured in centimeters.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
centimeters (cm)
  Baseline: number analyzed (Participants) | 242 | 34 | 85
  Baseline | 171.7 (9.39) | 172.2 (10.67) | 171.7 (11.81)
  Year 1: number analyzed (Participants) | 176 | 21 | 54
  Year 1 | 171.9 (9.50) | 174.0 (10.01) | 170.6 (11.88)
  Year 2: number analyzed (Participants) | 160 | 23 | 49
  Year 2 | 172.0 (9.20) | 172.7 (9.90) | 171.4 (12.13)
  Year 3: number analyzed (Participants) | 122 | 18 | 47
  Year 3 | 172.1 (9.68) | 172.5 (10.45) | 172.8 (11.54)
  Year 4: number analyzed (Participants) | 85 | 8 | 30
  Year 4 | 173.0 (9.40) | 172.5 (7.95) | 172.0 (11.60)
  Year 5: number analyzed (Participants) | 16 | 0 | 2
  Year 5 | 171.0 (11.44) |  | 169.1 (5.80)

9. Secondary Outcome: Change From Baseline in Height of Participants at Years 1, 2, 3, 4 and 5
Description: Height of participants was measured in centimeters.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
centimeters (cm)
  Change at Year 1: number analyzed (Participants) | 174 | 21 | 53
  Change at Year 1 | 0 (0.31) | -0.1 (0.78) | 0 (0.31)
  Change at Year 2: number analyzed (Participants) | 156 | 21 | 49
  Change at Year 2 | 0 (0.30) | -0.1 (0.79) | 0 (0.17)
  Change at Year 3: number analyzed (Participants) | 119 | 15 | 46
  Change at Year 3 | 0 (0.60) | 0 (0) | 0 (0.35)
  Change at Year 4: number analyzed (Participants) | 84 | 6 | 30
  Change at Year 4 | 0 (0.56) | 0 (0) | 0 (0.21)
  Change at Year 5: number analyzed (Participants) | 15 | 0 | 2
  Change at Year 5 | -0.1 (0.52) |  | 0 (0)

10. Secondary Outcome: Body Mass Index (BMI) of Participants at Baseline, Years 1, 2, 3, 4 and 5
Description: BMI was defined as an index for assessing overweight and underweight and was obtained by dividing body weight in kilograms (kg) by height in meters squared (m^2).
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kilogram per meter squared (kg/m^2)
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
Kilogram per meter squared (kg/m^2)
  Baseline: number analyzed (Participants) | 231 | 31 | 80
  Baseline | 28.3 (4.76) | 27.8 (5.71) | 29.6 (8.42)
  Year 1: number analyzed (Participants) | 168 | 19 | 51
  Year 1 | 28.2 (5.45) | 28.3 (5.56) | 28.9 (7.26)
  Year 2: number analyzed (Participants) | 156 | 20 | 45
  Year 2 | 27.9 (4.20) | 28.9 (4.70) | 29.8 (6.08)
  Year 3: number analyzed (Participants) | 102 | 14 | 45
  Year 3 | 28.8 (5.55) | 28.5 (4.70) | 29.8 (6.47)
  Year 4: number analyzed (Participants) | 70 | 5 | 27
  Year 4 | 27.4 (4.09) | 33.2 (2.92) | 28.2 (7.24)
  Year 5: number analyzed (Participants) | 11 | 0 | 2
  Year 5 | 27.8 (6.14) |  | 36.6 (2.81)

11. Secondary Outcome: Change From Baseline in Body Mass Index of Participants at Years 1, 2, 3, 4 and 5
Description: BMI was defined as an index for assessing overweight and underweight and was obtained by dividing body weight in kilograms (kg) by height in m^2.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
kg/m^2
  Change at Year 1: number analyzed (Participants) | 162 | 17 | 49
  Change at Year 1 | 0 (2.67) | -0.4 (4.60) | -0.9 (7.79)
  Change at Year 2: number analyzed (Participants) | 149 | 17 | 45
  Change at Year 2 | -0.2 (2.25) | -0.5 (3.84) | 0.3 (2.03)
  Change at Year 3: number analyzed (Participants) | 97 | 12 | 39
  Change at Year 3 | 0.7 (3.75) | -0.3 (4.13) | -1.1 (6.02)
  Change at Year 4: number analyzed (Participants) | 66 | 4 | 26
  Change at Year 4 | -0.4 (2.62) | 1.8 (2.43) | -0.1 (2.54)
  Change at Year 5: number analyzed (Participants) | 11 | 0 | 2
  Change at Year 5 | -0.7 (2.85) |  | -4.3 (6.78)

12. Secondary Outcome: Blood Pressure (BP) of Participants at Baseline, Years 1, 2, 3, 4 and 5
Description: Measurement of BP included supine systolic blood pressure (SBP) and diastolic blood pressure (DBP).
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
millimeter of mercury (mmHg)
  Supine SBP- Baseline: number analyzed (Participants) | 227 | 35 | 69
  Supine SBP- Baseline | 132.3 (16.47) | 123.6 (13.47) | 120.3 (13.40)
  Supine SBP- Year 1: number analyzed (Participants) | 171 | 20 | 51
  Supine SBP- Year 1 | 132.7 (17.82) | 127.4 (16.00) | 122.9 (11.74)
  Supine SBP- Year 2: number analyzed (Participants) | 161 | 21 | 47
  Supine SBP- Year 2 | 133.3 (16.82) | 133.5 (21.97) | 124.1 (14.37)
  Supine SBP- Year 3: number analyzed (Participants) | 114 | 16 | 45
  Supine SBP- Year 3 | 133.4 (15.68) | 130.4 (20.13) | 123.4 (14.26)
  Supine SBP- Year 4: number analyzed (Participants) | 77 | 7 | 29
  Supine SBP- Year 4 | 132.3 (14.80) | 134.4 (14.01) | 127.8 (13.97)
  Supine SBP- Year 5: number analyzed (Participants) | 14 | 0 | 2
  Supine SBP- Year 5 | 137.4 (17.76) |  | 121.0 (1.41)
  Supine DBP- Baseline: number analyzed (Participants) | 227 | 35 | 69
  Supine DBP- Baseline | 78.4 (9.32) | 75.5 (10.76) | 74.0 (8.29)
  Supine DBP- Year 1: number analyzed (Participants) | 171 | 20 | 51
  Supine DBP- Year 1 | 77.1 (9.37) | 73.0 (11.00) | 74.6 (9.01)
  Supine DBP- Year 2: number analyzed (Participants) | 161 | 21 | 47
  Supine DBP- Year 2 | 78.2 (9.10) | 75.8 (12.32) | 76.3 (9.06)
  Supine DBP- Year 3: number analyzed (Participants) | 114 | 16 | 45
  Supine DBP- Year 3 | 79.0 (9.04) | 77.2 (10.99) | 76.0 (7.84)
  Supine DBP- Year 4: number analyzed (Participants) | 77 | 7 | 29
  Supine DBP- Year 4 | 77.5 (9.01) | 80.6 (11.91) | 76.1 (8.04)
  Supine DBP- Year 5: number analyzed (Participants) | 14 | 0 | 2
  Supine DBP- Year 5 | 80.6 (12.82) |  | 70.5 (0.71)

13. Secondary Outcome: Change From Baseline in Blood Pressure of Participants at Years 1, 2, 3, 4 and 5
Description: Measurement of BP included supine SBP and DBP.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
mmHg
  Change in Supine SBP- Year 1: number analyzed (Participants) | 161 | 19 | 40
  Change in Supine SBP- Year 1 | 1.0 (15.67) | -0.9 (11.52) | 3.4 (13.52)
  Change in Supine SBP- Year 2: number analyzed (Participants) | 152 | 18 | 37
  Change in Supine SBP- Year 2 | 0.4 (15.78) | 6.1 (17.48) | 2.3 (12.81)
  Change in Supine SBP- Year 3: number analyzed (Participants) | 105 | 14 | 32
  Change in Supine SBP- Year 3 | 1.0 (13.84) | 1.5 (17.11) | 4.3 (12.41)
  Change in Supine SBP- Year 4: number analyzed (Participants) | 71 | 6 | 22
  Change in Supine SBP- Year 4 | -1.5 (19.91) | 10.5 (10.65) | 4.3 (16.40)
  Change in Supine SBP- Year 5: number analyzed (Participants) | 14 | 0 | 2
  Change in Supine SBP- Year 5 | 5.7 (19.26) |  | -4.0 (8.49)
  Change in Supine DBP- Year 1: number analyzed (Participants) | 161 | 19 | 40
  Change in Supine DBP- Year 1 | -1.2 (10.66) | -4.2 (10.2) | 0.6 (9.83)
  Change in Supine DBP- Year 2: number analyzed (Participants) | 152 | 18 | 37
  Change in Supine DBP- Year 2 | -0.6 (10.84) | 0.5 (11.81) | 1.8 (8.17)
  Change in Supine DBP- Year 3: number analyzed (Participants) | 105 | 14 | 32
  Change in Supine DBP- Year 3 | 0.7 (10.44) | -0.4 (8.2) | 0.8 (8.81)
  Change in Supine DBP- Year 4: number analyzed (Participants) | 71 | 6 | 22
  Change in Supine DBP- Year 4 | -1.5 (12.07) | -2.8 (9.77) | 2.0 (9.50)
  Change in Supine DBP- Year 5: number analyzed (Participants) | 14 | 0 | 2
  Change in Supine DBP- Year 5 | 3.0 (12.36) |  | 0.5 (0.71)

14. Secondary Outcome: Heart Rate of Participants at Baseline, Years 1, 2, 3, 4 and 5
Description: Heart rate was measured in supine position.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
beats per minute (bpm)
  Baseline: number analyzed (Participants) | 169 | 30 | 50
  Baseline | 69.3 (9.42) | 68.7 (10.66) | 69.7 (8.28)
  Year 1: number analyzed (Participants) | 137 | 18 | 41
  Year 1 | 70.2 (11.22) | 70.7 (13.39) | 74.1 (10.79)
  Year 2: number analyzed (Participants) | 129 | 18 | 33
  Year 2 | 69.8 (10.41) | 70.5 (14.46) | 71.3 (11.05)
  Year 3: number analyzed (Participants) | 84 | 14 | 35
  Year 3 | 71.5 (9.90) | 69.8 (10.59) | 69.0 (11.08)
  Year 4: number analyzed (Participants) | 58 | 6 | 25
  Year 4 | 68.3 (9.15) | 64.3 (15.34) | 69.4 (11.68)
  Year 5: number analyzed (Participants) | 11 | 0 | 1
  Year 5 | 68.5 (10.92) |  | 70.0 (NA) — Standard deviation was not estimable because only 1 participant was analyzed.

15. Secondary Outcome: Change From Baseline in Heart Rate of Participants at Years 1, 2, 3, 4 and 5
Description: Heart rate was measured in supine position.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
bpm
  Change at Year 1: number analyzed (Participants) | 113 | 16 | 26
  Change at Year 1 | 1.4 (11.62) | -1.4 (12.66) | 4.7 (12.06)
  Change at Year 2: number analyzed (Participants) | 100 | 13 | 24
  Change at Year 2 | 0.7 (10.57) | 1.8 (14.88) | 3.4 (11.47)
  Change at Year 3: number analyzed (Participants) | 65 | 10 | 18
  Change at Year 3 | 0.1 (13.24) | 1.5 (13.94) | 1.6 (15.11)
  Change at Year 4: number analyzed (Participants) | 44 | 4 | 15
  Change at Year 4 | 1.3 (8.97) | 1.0 (16.31) | 0.7 (9.76)
  Change at Year 5: number analyzed (Participants) | 9 | 0 | 1
  Change at Year 5 | 3.7 (13.49) |  | 0 (NA) — Standard deviation was not estimable because only 1 participant was analyzed.

16. Secondary Outcome: Percentage of Participants With Body Composition Assessments at Baseline, Years 1, 2, 3 and 4
Description: Body composition included parameters fat mass and muscle mass.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
percentage of participants
  Baseline | 48.78 | 47.37 | 58.62
  Year 1 | 31.30 | 5.26 | 31.03
  Year 2 | 33.33 | 21.05 | 34.48
  Year 3 | 15.85 | 21.05 | 20.69
  Year 4: number analyzed (Participants) | 246 | 0 | 87
  Year 4 | 2.03 |  | 5.75

17. Secondary Outcome: Percentage of Participants With Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) Investigation at Baseline, Years 1, 2, 3, 4 and 5
Description: CT is a diagnostic imaging test used to create detailed images of internal organs, bones, soft tissue and blood vessels. MRI investigation uses strong magnetic field and radio waves to create detailed images of the organs and tissues within the body.
Time Frame: Baseline, Year 1, 2, 3, 4, 5
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
percentage of participants
  Baseline | 32.93 | 42.11 | 18.39
  Year 1 | 14.63 | 23.68 | 6.9
  Year 2 | 15.04 | 13.16 | 3.45
  Year 3 | 11.38 | 7.89 | 5.75
  Year 4 | 4.88 | 5.26 | 4.6
  Year 5: number analyzed (Participants) | 246 | 0 | 87
  Year 5 | 1.63 |  | 1.15

18. Secondary Outcome: Percentage of Participants With Any Change From Baseline in Hormone Abnormalities at Years 1, 2, 3, and 4
Description: Hormones that were evaluated were thyroid stimulating hormone, adrenocorticotropic hormone, luteinizing hormone, follicle-stimulating hormone, antidiuretic hormone and prolactin hormone. Abnormalities were judged by the investigator.
Time Frame: Baseline, Year 1, 2, 3, 4
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 246 | 38 | 87
percentage of participants
  Year 1 | 2.03 | 2.63 | 1.15
  Year 2: number analyzed (Participants) | 246 | 0 | 87
  Year 2 | 1.63 |  | 1.15
  Year 3 | 1.63 | 2.63 | 1.15
  Year 4: number analyzed (Participants) | 246 | 38 | 0
  Year 4 | 0.41 | 2.63 |

19. Secondary Outcome: Percentage of Participants With Any Concomitant Medication at Baseline and During Follow-up
Description: Percentage of participants taking any medications other than Genotropin (concomitant medication) are reported.
Time Frame: Baseline, Follow-up (during 28 days after last dose of Genotropin treatment)
Population: All participants who were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
Number analyzed (Participants) | 247 | 42 | 88
percentage of participants
  Baseline | 83.0 | 69.0 | 83.0
  During follow-up | 92.3 | 73.8 | 88.6

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of Genotropin treatment (maximum up to 5 years)
Description: Same event may appear as an AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study. Participants treated with at least 1 dose of Genotropin were evaluated for safety.
Arm/Group | KIMS Adult Onset Growth Hormone Deficiency (GHD) | Naive Adult Onset GHD | Childhood Onset Growth Hormone Deficiency (CO-GHD)
All-Cause Mortality (participants affected / at risk) | 12/246 | 1/41 | 0/87
Serious Adverse Events (participants affected / at risk) | 57/246 | 5/41 | 10/87
Other Adverse Events (participants affected / at risk) | 66/246 | 14/41 | 15/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KIMS Adult Onset Growth Hormone Deficiency (GHD) (N=246) | Naive Adult Onset GHD (N=41) | Childhood Onset Growth Hormone Deficiency (CO-GHD) (N=87)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pituitary tumour recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Guillain-barre syndrome (Nervous system disorders) | 0 | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0
Cortisol deficiency (Endocrine disorders) | 0 | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 1 | 0 | 0
Hyperparat hyroidism (Endocrine disorders) | 1 | 0 | 0
Pituitary apoplexy (Endocrine disorders) | 1 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Dysplasia (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0
Strangulated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Neurofibromatosis (Congenital, familial and genetic disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Amputation (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KIMS Adult Onset Growth Hormone Deficiency (GHD) (N=246) | Naive Adult Onset GHD (N=41) | Childhood Onset Growth Hormone Deficiency (CO-GHD) (N=87)
Headache (Nervous system disorders) | 1 | 3 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 0
Visual field defect (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 1
Dementia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Upper respiratory track infection (Infections and infestations) | 2 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 0 | 0
Malaria (Infections and infestations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fatigue (General disorders) | 7 | 2 | 2
Pyrexia (General disorders) | 2 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Prostatic specific antigen increased (Investigations) | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Colonoscopy (Investigations) | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Blood prolactin increased (Investigations) | 1 | 0 | 0
Blood testosterone increased (Investigations) | 1 | 0 | 0
Blood homocysteine increased (Investigations) | 1 | 0 | 0
Blood folate decreased (Investigations) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Aneurysm (Vascular disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 1
Libido decreased (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 3 | 0 | 0
Hyperparat hyroidism primary (Endocrine disorders) | 1 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 2 | 0 | 0
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 1
Gastric banding (Surgical and medical procedures) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1
Syringe issue (Product Issues) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-10-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT01947894/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT01947894/SAP_001.pdf